CLINICAL TRIAL: NCT02204488
Title: Total Joint Arthroplasty or Trapeziectomy for Treating Trapeziometacarpal Osteoarthritis Eaton & Glickel Stage 2 and 3: a Randomized Clinical Trial
Brief Title: Surgical Treatment for Trapeziometacarpal Osteoarthritis Eaton & Glickel Stage 2-3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Isala (Other)
Responsible Party: Principal Investigator, Ramon de Wildt, MD, Isala
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NL47755.075.14; NL47755.075.14 (Registry Identifier: METC Isala)
Record Dates: First submitted 2014-07-29; First posted 2014-07-30 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Trapeziometacarpal Osteoarthritis; Thumb Carpometacarpal Osteoarthritis
Keywords: Osteoarthritis; Thumb; Total joint arthroplasty; Trapeziectomy
MeSH Terms: conditions — Osteoarthritis | interventions — Arthroplasty, Replacement

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Joint Arthroplasty (Active Comparator): Total Joint Arthroplasty
  Interventions: Procedure: Total Joint Arthroplasty
- Trapeziectomy (Active Comparator): Trapeziectomy
  Interventions: Procedure: Trapeziectomy

INTERVENTIONS:
Procedure: Total Joint Arthroplasty — Total Joint Arthroplasty with device: Maïa® trapezio-metacarpal joint prosthesis, Groupe Lépine, Genay, France
  Arms: Total Joint Arthroplasty
Procedure: Trapeziectomy — Trapeziectomy
  Arms: Trapeziectomy

SUMMARY:
Trapeziometacarpal osteoarthritis is a common cause of pain and loss of hand function in postmenopausal women. Many surgical treatments have been described and recent literature has show that the relatively simple trapeziectomy gives equal results and less complications, when compared to other techniques such as ligament reconstructions and interpositions. A relatively new treatment modality, which has been further developed in recent years is the total joint arthroplasty. Randomized prospective trials and long-term results are lacking, but prospective cohorts show a faster recovery and good results after one year, without an increase in complication rate.

We hypothesize that a total joint arthroplasty gives a better objective and subjective result after one year than a trapeziectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women.
* 40 years of age or more.
* Symptomatic trapeziometacarpal osteoarthritis.
* Eaton & Glickel stage 2 and 3.

Exclusion Criteria:

* An operation for trapeziometacarpal osteoarthritis on the same hand in the past.
* Participation in randomized clinical trial for trapeziometacarpal osteoarthritis with contralateral hand.
* Secondary trapeziometacarpal osteoarthritis as result of trauma, rheumatoid arthritis, systemic lupus or gout.
* Symptomatic carpal tunnel syndrome in same hand.
* Symptomatic Quervain's tenosynovitis in same hand.
* Neurological or other disorders of the affected side that can influence postoperative rehabilitation.
* Insufficient knowledge of Dutch language.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Michigan Hand Outcomes Questionnaire (MHOQ) | 1 year after surgery
  Is there a difference is daily hand function between patients with a total joint arthroplasty and patients with a trapeziectomy after 1 year postoperatively, measured with the total score of the Michigan Hand Outcomes Questionnaire (MHOQ)?

SECONDARY OUTCOMES:
Michigan Hand Outcomes Questionnaire (MHOQ) | 5 years after surgery
  Is there a difference is daily hand function between patients with a total joint arthroplasty and patients with a trapeziectomy after 5 years postoperatively, measured with the total score of the Michigan Hand Outcomes Questionnaire (MHOQ)?
Michigan Hand Outcomes Questionnaire (MHOQ) | 1 and 5 years after surgery
  Is there a difference is daily hand function between patients with a total joint arthroplasty and patients with a trapeziectomy after 1 and 5 years postoperatively, measured with the different subscales (i.e. pain) of the Michigan Hand Outcomes Questionnaire (MHOQ)?
Disabilities of Arm Shoulder and Hand (DASH) | 1 and 5 years after surgery
  Is there a difference is daily hand function after 1 and 5 years postoperatively between patients with a total joint arthroplasty and patients with a trapeziectomy measured with the Disabilities of Arm Shoulder and Hand (DASH)?
Grip strength | 1 and 5 years after surgery
  Is there a difference in grip strength between patients with a total joint arthroplasty and patients with a trapeziectomy after 1 and 5 years?
Thumb mobility | 1 and 5 years after surgery
  Is there a difference in mobility of the thumb between patients with a total joint arthroplasty and patients with a trapeziectomy after 1 and 5 years?
Complications | 1 and 5 years after surgery
  Is there a difference in postoperative complications between patients with a total joint arthroplasty and patients with a trapeziectomy after 1 and 5 years?
Return to work | 1 and 5 years after surgery
  Is there a difference in return to work between patients with a total joint arthroplasty and patients with a trapeziectomy after 1 and 5 years?

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen H. van Uchelen, MD, Study Director — Isala
Locations (1):
- Isala Hospital, Zwolle, Overijssel, Netherlands